CLINICAL TRIAL: NCT05289479
Title: Effect Of Repeated Pre-Heating Of Resin Composite Restoration On Its Clinical Performance And Post-Operative Dentin Hypersensitivity "A Randomized Clinical Trial"
Brief Title: Pre-heated Resin Composite Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Elkady, Assistant Lecturer at Department of Conservative Dentistry, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 73-11\9\2022-440
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: The Effect of Preheating Cycles of Resin Composite on Both Hypersensitivity and Clinical Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No pre-heating "control group" (Active Comparator): resin composite is used at room temperature without preheating
  Interventions: Procedure: no pre-heating of resin composite before application
- 0ne cycle pre-heating (Active Comparator): one cycle preheating of resin composite at 68 degree Celsius before application
  Interventions: Procedure: Pre-heating of resin composite before application
- ten cycles pre-heating (Active Comparator): ten cycles preheating of resin composite at 68 degree Celsius before application
  Interventions: Procedure: Pre-heating of resin composite before application

INTERVENTIONS:
Procedure: Pre-heating of resin composite before application — the effect of preheating of resin composite before application in class II cavities
  Arms: 0ne cycle pre-heating; ten cycles pre-heating
Procedure: no pre-heating of resin composite before application — The control group
  Arms: No pre-heating "control group"

SUMMARY:
this study is conducted to evaluate the post-operative hypersensitivity and clinical performance of preheated resin composite with different number of pre-heating cycles in class II carious lesions compared to resin composite restorations without preheating using Modified US Public Health Service Clinical Criteria (USPHS).

DETAILED DESCRIPTION:
1. Scientific Background One of the main problems associated with composite resin restorations is poor adaptation and gap formation between the restorative material and the cavity walls, resulting in the micro-leakage of oral fluids and accumulation of fluids responsible for many problems such as postoperative hypersensitivity, marginal discoloration and recurrent caries.

   Despite of recent developments in dental restorative materials and techniques, postoperative sensitivity following the application of a posterior resin composite restoration is often reported by dentists, as a clinical problem.

   Pre-application warming of dental resin composite restorative materials, is considered one of the modern modifications for the application of resin composite, which reduces viscosity and increases flowability, that in turn secures superior adaptation to the prepared cavity walls.

   Resin composite warming appliances found in the market nowadays, offer multiple choices for preheating either in different temperatures or in the form of the cassettes which could be compatible with different supplied forms from different manufacturers "capsules or syringes". Multiple cycles of preheating for the used composite resin syringe can affect both marginal integrity and mechanical properties of the resin composite according to the number of cycles applied.

   Increasing the temperature of dental resin composite before application can aid in monomer mobility inside its matrix giving high quality of degree of conversion and more highly cross-linked polymeric network. This kind of change of the rheology of the resin composite can aid in decreasing the postoperative hyper-sensitivity.

   However, an intensive review of literature failed to disclose the effect of using resin composite preheated for multiple times with different temperatures on the post-operative hypersensitivity.
2. Statement of the problem Using the same resin composite syringe that previously preheated multiple times in different daily restorative cases, can adversely affect the properties and the performance of the applied resin composite.
3. Hypothesis The null hypothesis is that using resin composite previously preheated for different cycles will not be different in reducing postoperative hypersensitivity, marginal integrity and mechanical properties of the resin composite as without preheating.

D. The sample size calculation

1. primary outcome: This power analysis used marginal integrity after 12 months as the primary outcome. Based upon the results of Kurdi R and Abboud SA (2016); Bulk Fill composite showed 13 cases with (Alpha) score and 4 cases with (Beta) score, respectively. The effect size (w) was 0.53. Using alpha (α) level of (5%) and Beta (β) level of (20%) i.e. power = 80%; the minimum estimated sample size was 28 cases. Sample size was increased to 35 cases to compensate for a drop-out rate of 25% after 12 months. Sample size calculation was performed using G*Power Version 3.1.9.2.
2. secondary outcome: This power analysis used hypersensitivity grades after one day in patient with medium cavity depth as the primary outcome. The effect sizes w1 = (1.4) and w2 = (1.11) were calculated based upon the results of Ragab H (2018). Using alpha (α) level of (5%) and Beta (β) level of (20%) i.e. power = 80%; the minimum estimated sample size was a total of 11 subjects. Sample size was increased to a total of 14 subjects (7 subjects per group) to compensate for a dropout rate of 25%. Sample size calculation was performed using G*Power Version 3.1.9.2

ELIGIBILITY:
Inclusion Criteria:

* 1- Moderate to deep proximal primary carious lesions" Class II" where each patient will have 2 "Class II" cavities on different sides.

  2- Overall good oral hygiene status 3- Patients showing no signs of spontaneous dental or orofacial pain. 4- Selected teeth should not have any signs or symptoms of pulpal and periapical disease.

  5- The selected teeth should have an occlusal contact with natural or crowned antagonist teeth, so that it could be tested for post-operative pain during chewing of food.

  6- The selected teeth should have healthy gingival tissues, without gingival recession or alveolar bone loss.

Exclusion Criteria:

* 1. Patients with a compromised medical history, or had received therapeutic irradiation to the head and neck region.

  2. Acute and chronic systemic diseases, immune-compromised patients. 3. Medical problems preventing the participant from showing up to describe the presence of hypersensitivity 4. Alcoholic and smoker patients. 5. Pregnant or breastfeeding 6. Patients having physical disabilities, or who are unable to brush their teeth 7. Patients who have a history of allergies to any personal oral care product or ingredient, or who are taking anti-inflammatory drugs within the previous month.

  8. Patients taking analgesics that could alter their normal pain perception level.

  9. Medical, psychiatric, or pharmaco-therapeutic histories that might compromise the study protocol including chronic use of ant-inflammatory, analgesic, psychotropic drugs.

  10. Individuals who had sensitive teeth but with one of the following conditions will be excluded from the study, teeth with large restorations, abutment of teeth of removable par¬tial dentures, dental caries, enamel cracks, leakage of fillings or other restorations, cracked teeth, dental pulp lesions, den¬tal abscesses, pulpitis, and atypical facial pain.

  11. Defective restorations that needs replacement for esthetic reasons. 12. Patient with severe periodontitis or severe erosion damage. 13. Patients had participated in a clinical trial within 6 months before commencement of this trial.

  14. Patients unable to return for recall appointment. 15. Previously restored teeth showing secondary caries. 16. Occlusal disturbances or temporo-mandibular joint problems involving gingival recession or alveolar bone loss.

  17. Patients on orthodontic treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
United States Public Health Service (USPHS) criteria | 9 months
  Clinical performance of the restorations tested for 9 months

SECONDARY OUTCOMES:
Post-Operative Dentin Hypersensitivity | 1 month
  Intensity of postoperative pain measured using a Modified Visual Analogue scale before and after filling for 1 month postoperatively.
  The score of scale from 0 to 10 where zero has no postoperative sensitivity at all and ten means the worst postoperative sensitivity is felt by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minya, Minia City, Egypt